CLINICAL TRIAL: NCT01827735
Title: Adaptive Study of IL-2 Dose on Regulatory T Cells in Type 1 Diabetes (DILT1D)
Brief Title: Regulatory T Cells in Type 1 Diabetes Patients Treated With IL-2
Acronym: DILT1D
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Juvenile Diabetes Research Foundation (Other); National Institute for Health Research, United Kingdom (Other Government); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Dr Frank Waldron-Lynch, Academic Consultant Endocrinologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A092737; ISRCTN27852285 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2013-04-04; First posted 2013-04-10 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Type 1 Diabetes
Keywords: Interleukin 2; Type 1 diabetes; T regulatory cells; Adaptive trial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aldesleukin (Proleukin) — A single, subcutaneous dose will be given administered with the maximum dose allowed 1.5 X 106 IU/M2.

SUMMARY:
Type 1 diabetes is the most common severe chronic autoimmune disease worldwide and is caused by the autoimmune (loss of self tolerance) mediated destruction of the insulin producing pancreatic beta cells thus leading to insulin deficiency and development of hyperglycaemia. Currently, medical management of type 1 diabetes focuses on intensive insulin replacement therapy to limit complications (retinopathy, nephropathy, neuropathy); nevertheless clinical outcomes remain sub optimal. There are intensive efforts to design novel immunotherapies that can arrest the autoimmune process and thereby preserve residual insulin production leading to fewer complications and better clinical outcomes.

The vast majority of genes that contribute to susceptibility to type 1 diabetes have been found to encode proteins involved in immune regulation and function. In particular, several susceptibility proteins are involved in the interleukin 2 (IL-2) pathway that regulates T cell activation and tolerance to self antigens. Aldesleukin is a human recombinant IL-2 product produced by recombinant DNA technology using genetically engineered E. coli stain containing an analog of the human interleukin-2 gene. There is substantial nonclinical, preclinical and clinical data that ultra low dose IL-2 (aldesleukin) therapy can arrest the autoimmune mediated destruction of pancreatic beta cells by induction of functional T regulatory cells. However, prior to embarking on large proof of concept trials in type 1 diabetes it is essential that the optimum dose of IL-2 (aldesleukin) is determined. The objective of this study is to establish in patients with type 1 diabetes the optimal dose of IL-2 (aldesleukin) to administer in order to increase T regulatory cell response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Type 1 diabetes
* 18-50 years
* Duration of diabetes less than 24 months from diagnosis
* One positive autoantibody (anti-islet cell, anti-GAD, anti-IA2, anti-ZnT8)

Exclusion Criteria:

* Hypersensitivity to aldesleukin or any of the excipients
* History of severe cardiac disease
* History of malignancy within the past 5 years (with the exception of localized carcinoma of the skin that had been resected for cure or cervical carcinoma in situ)
* History or concurrent use of immunosuppressive agents or steroids
* History of unstable diabetes with recurrent hypoglycaemia
* Active autoimmune, hyper or hypothyroidism
* Active clinical infection
* Major pre-existing organ dysfunction or previous organ allograft
* Females who are pregnant, lactating or intend to get pregnant during the study - Males who intend to father a pregnancy during the study
* Donation of more than 500 ml of blood within 2 months prior to aldesleukin administration
* Participation in a previous therapeutic clinical trial within 2 months prior to aldesleukin administration
* Abnormal ECG Abnormal full blood count, chronic renal failure (Stage 3,4,5) and/or evidence impaired liver function
* Positive Hepatitis B surface Antigen (HBsAg) or Hepatitis C serology or Human Immunodeficiency Virus (HIV) test
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the patient ineligible for inclusion because of a safety concern

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is based upon the percentage of CD4+T regulatory (defined as CD3+CD4+CD25highCD127low) cells within the CD3+CD4+T cell gate following treatment with IL-2. | From Day 0 to Day 60
  Fluorescence-activated cell sorting assay

SECONDARY OUTCOMES:
T regulatory cell phenotype and stability | From Day 0 to Day 60
  Fluorescence-activated cell sorting assay
T effector cell number and phenotype | From Day 0 - Day 60
  Fluorescence-activated cell sorting assay
T cell subset proliferation and populations | From Day 0 - Day 60
  Fluorescence-activated cell sorting assay
Intracellular T cell and natural killer(NK) cell signalling | From Day 0 - Day 60
  Fluorescence-activated cell sorting assay
T regulatory cell function | From Day 0 - Day 60
  T suppression assay
IL-2 pathway genotype | From Day 0 - Day 60
  DNA sequencing
Lymphocyte Subsets | From Day 0 to Day 60
  Complete blood count
Serum Cytokines | From Day 0 to Day 60
  Enzyme-linked immuno sorbent assay
Glycaemic control | From Day 0 to Day 60
  Self monitoring blood glucose readings, HbA1c, insulin usage
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | From Day O to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Frank Waldron-Lynch, Principal Investigator — University of Cambridge
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrooke's Hospital, Cambridge, United Kingdom

REFERENCES:
- [Background] Waldron-Lynch F, Kareclas P, Irons K, Walker NM, Mander A, Wicker LS, Todd JA, Bond S. Rationale and study design of the Adaptive study of IL-2 dose on regulatory T cells in type 1 diabetes (DILT1D): a non-randomised, open label, adaptive dose finding trial. BMJ Open. 2014 Jun 4;4(6):e005559. doi: 10.1136/bmjopen-2014-005559. PMID 24898091
- [Result] Heywood J, Evangelou M, Goymer D, Kennet J, Anselmiova K, Guy C, O'Brien C, Nutland S, Brown J, Walker NM, Todd JA, Waldron-Lynch F. Effective recruitment of participants to a phase I study using the internet and publicity releases through charities and patient organisations: analysis of the adaptive study of IL-2 dose on regulatory T cells in type 1 diabetes (DILT1D). Trials. 2015 Mar 11;16:86. doi: 10.1186/s13063-015-0583-7. PMID 25881192
- [Derived] Todd JA, Evangelou M, Cutler AJ, Pekalski ML, Walker NM, Stevens HE, Porter L, Smyth DJ, Rainbow DB, Ferreira RC, Esposito L, Hunter KM, Loudon K, Irons K, Yang JH, Bell CJ, Schuilenburg H, Heywood J, Challis B, Neupane S, Clarke P, Coleman G, Dawson S, Goymer D, Anselmiova K, Kennet J, Brown J, Caddy SL, Lu J, Greatorex J, Goodfellow I, Wallace C, Tree TI, Evans M, Mander AP, Bond S, Wicker LS, Waldron-Lynch F. Regulatory T Cell Responses in Participants with Type 1 Diabetes after a Single Dose of Interleukin-2: A Non-Randomised, Open Label, Adaptive Dose-Finding Trial. PLoS Med. 2016 Oct 11;13(10):e1002139. doi: 10.1371/journal.pmed.1002139. eCollection 2016 Oct. PMID 27727279
- See also: DILT1D trial facebook page — https://www.facebook.com/ClinicalTrialsType1Diabetes
- See also: DILT1D trial Twitter update — https://twitter.com/t1diabetestrial